CLINICAL TRIAL: NCT06116539
Title: Multicenter Randomized Clinical Trial of the Use of Cyanoacrylate in Healing and Pain in the Palatal Donor Site of Connective Tissue Grafts
Brief Title: Use of Cyanoacrylate in Healing and Pain in the Palatal Donor Site of Connective Tissue Grafts
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alfonso X El Sabio University (Other)
Responsible Party: Principal Investigator, Joaquin Lopez-Malla, Master on Oral Surgery, Implantology and Periodontic´s professor, Alfonso X El Sabio University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: cyanoacrylate multicenter
Record Dates: First submitted 2023-09-18; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-09

CONDITIONS: Pain, Postoperative; Healing Surgical Wounds
Keywords: tissue adhesive; wound dressing; cyanoacrylate; gingival graft; palatal graft; conective tissue graft
MeSH Terms: conditions — Pain, Postoperative | interventions — Cyanoacrylates; Sutures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cyanoacrylate Group (Experimental): In the test group, a cyanoacrylate-based tissue adhesive (PeriAcryl 90 HV; Glustitch, Delta, Canada) will be applied.
  Interventions: Drug: Cyanoacrylate
- Suture Group (Active Comparator): In the control group, the edges will be approximated with 4/0 monofilament non-absorbable nylon suture (Aragó, Barcelona, Spain).
  Interventions: Procedure: Suture

INTERVENTIONS:
Drug: Cyanoacrylate — In the test group, a cyanoacrylate-based tissue adhesive (PeriAcryl 90 HV; Glustitch, Delta, Canada) will be applied.
  Arms: Cyanoacrylate Group
Procedure: Suture — After harvesting the full-thickness connective tissue graft, the edges of the control group will be approximated with 4/0 non-absorbable monofilament nylon suture (Aragó, Barcelona, Spain).
  Arms: Suture Group

SUMMARY:
Periodontal plastic surgery has been performed successfully for a long time in the treatment of gingival recessions and mucogingival defects. Epithelial and connective tissue grafts are considered the "gold standard" treatment for gingival recession due to their biocompatibility and long-term stability, however they require tissue harvesting from a donor area, usually the palate, increasing patient discomfort. Various hemostatic and healing agents have been used in conjunction with suturing to speed healing and reduce complications associated with this procedure, such as bleeding and pain. These include absorbable synthetic collagen, absorbable gelatin sponges, oxidized regenerated cellulose, ferric subsulfate, and more recently, cyanoacrylate cements and platelet-rich fibrin. Cyanoacrylate adhesives are synthesized as monomers by condensation of a cyanoacetate with formaldehyde in the presence of catalysts and the adhesive film is developed by rapid polymerization caused by hydroxide groups to the surfaces to be adhered. The properties of cyanoacrylate tissue adhesives of greatest interest in the surgical field are excellent hemostasis, rapid tissue adhesion, and possible bacteriostatic qualities.

DETAILED DESCRIPTION:
Periodontal plastic surgery has been performed successfully for a long time in the treatment of gingival recessions and mucogingival defects. Epithelial and connective tissue grafts are considered the "gold standard" treatment for gingival recession due to their biocompatibility and long-term stability, however they require tissue harvesting from a donor area, usually the palate, increasing patient discomfort. Various hemostatic and healing agents have been used in conjunction with suturing to speed healing and reduce complications associated with this procedure, such as bleeding and pain. These include absorbable synthetic collagen, absorbable gelatin sponges, oxidized regenerated cellulose, ferric subsulfate, and more recently, cyanoacrylate cements and platelet-rich fibrin. Cyanoacrylate adhesives are synthesized as monomers by condensation of a cyanoacetate with formaldehyde in the presence of catalysts and the adhesive film is developed by rapid polymerization caused by hydroxide groups to the surfaces to be adhered. The properties of cyanoacrylate tissue adhesives of greatest interest in the surgical field are excellent hemostasis, rapid tissue adhesion, and possible bacteriostatic qualities.

The objective of this study will be to evaluate the perception of pain by the patient in the postoperative period of procedures for taking connective grafts from the palate in which cyanoacrylate-based tissue adhesive (PeriAcryl 90 HV; Glustitch, Delta, Canada) is used in comparison with a control group in which the clot was stabilized with the use of sutures.

Secondary Objectives:

To evaluate the healing of the palate in those patients in whom cyanoacrylate-based tissue adhesive (PeriAcryl 90 HV; Glustitch, Delta, Canada) is used, and compare it with a control group in which the clot is stabilized with the use of suture.

Evaluate the appearance of complications in procedures for taking connective grafts from the palate, such as necrosis or bleeding.

To evaluate the relationship between the dimensions of the connective tissue graft/thickness of the remaining epithelium after taking the graft and the appearance of complications.

Evaluate the time of the procedure in the harvesting of the graft, both in the suture and cyanoacrylate groups.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be considered a candidate for mucogingival treatment
* Requiring grafting around teeth or implants.
* No age limit is established for the sample.

Exclusion Criteria:

* Patients with systemic or scarring compromises
* Treated with bisphosphonates
* Smokers of more than 10 cigarettes a day
* With a history of previous palatal grafting in that location
* Present any type of contraindication to undergo surgery cannot take part in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Pain perception | Days 1,2,3,4,5,6,7 and 14 after the procedure
  The pain perceived by the patient will be evaluated by means of a Visual Analogue Scale (calibrated from 0 to 10, with 10 being the worst pain imaginable) during the first 1,2,3,4,5,6,7 and 14 days.

SECONDARY OUTCOMES:
Donor site healing | will be evaluated at 7 and 14 days after the procedure
  Donor site healing will be assessed visually at 7 and 14 days using the modified early wound healing index (MEHI),calibrated from 1 to 5, with 1 being complete closure with flap without a fibrin line on the palate, and 5 being incomplete closure of the flap with complete necrosis of the palatal tissue.

OTHER OUTCOMES:
intake of painkillers | 7 days after surgery
  Number of analgesics consumed during the first postoperative week

CONTACTS AND LOCATIONS:
Overall Officials: Joaquín LM Matute, dentistry, Study Director — Alfonso X El Sabio University
Locations (1):
- Joaquín López-Malla Matute, A Coruña, La Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alhourani MA, Kasem T, Hamadah O. Comparative study between using a tissue adhesive (N-BCA & OCA) and surgical sutures in free gingival graft surgery: A randomized controlled clinical trial. Dent Med Probl. 2022 Apr-Jun;59(2):241-248. doi: 10.17219/dmp/135382. PMID 35775864
- [Background] Basma HS, Saleh MHA, Abou-Arraj RV, Imbrogno M, Ravida A, Wang HL, Li P, Geurs N. Patient-reported outcomes of palatal donor site healing using four different wound dressing modalities following free epithelialized mucosal grafts: A four-arm randomized controlled clinical trial. J Periodontol. 2023 Jan;94(1):88-97. doi: 10.1002/JPER.22-0172. Epub 2022 Aug 3. PMID 35754198
- [Background] Castro-Gaspar C, Olmedo-Gaya MV, Romero-Olid MN, Lisbona-Gonzalez MJ, Vallecillo-Rivas M, Reyes-Botella C. Comparison between Tissue Adhesive Cyanoacrylate and Suture for Palatal Fibromucosa Healing: A Randomized Controlled Study. Materials (Basel). 2021 Nov 19;14(22):7009. doi: 10.3390/ma14227009. PMID 34832409
- [Background] Stavropoulou C, Atout RN, Brownlee M, Schroth RJ, Kelekis-Cholakis A. A randomized clinical trial of cyanoacrylate tissue adhesives in donor site of connective tissue grafts. J Periodontol. 2019 Jun;90(6):608-615. doi: 10.1002/JPER.18-0475. Epub 2018 Dec 26. PMID 30517975
- [Background] Tavelli L, Asa'ad F, Acunzo R, Pagni G, Consonni D, Rasperini G. Minimizing Patient Morbidity Following Palatal Gingival Harvesting: A Randomized Controlled Clinical Study. Int J Periodontics Restorative Dent. 2018 Nov/Dec;38(6):e127-e134. doi: 10.11607/prd.3581. PMID 30304077
- [Background] Tavelli L, Ravida A, Saleh MHA, Maska B, Del Amo FS, Rasperini G, Wang HL. Pain perception following epithelialized gingival graft harvesting: a randomized clinical trial. Clin Oral Investig. 2019 Jan;23(1):459-468. doi: 10.1007/s00784-018-2455-5. Epub 2018 Apr 30. PMID 29713890